CLINICAL TRIAL: NCT02678637
Title: Calf Muscle Strength in Patients Affected by Mitochondrial Diseases as Compared to Healthy Individuals
Brief Title: Calf Muscle Strength in Mitochondrial Diseases
Acronym: CMSMD
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Nanna Scharff Nielsen, Student researcher, Rigshospitalet, Denmark
Other Study IDs: H-1600058
Record Dates: First submitted 2016-02-03; First posted 2016-02-10 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Mitochondrial Disease
Keywords: MRI; CCSA; Contractile Cross Sectional Area; Strength; Calf muscle
MeSH Terms: conditions — Mitochondrial Diseases | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: MRI and muscle dynamometer

SUMMARY:
Mitochondrial disorders are a group of inherited disorders causing malfunctional mitochondria. Mitochondria are found in every cell of the body, and the disorders therefore give symptoms from every tissue, especially those with high energy needs as the brain, heart and muscles. The disorders are highly disabling.

The aim of the study is to investigate the relation between muscle strength and contractile cross sectional area (CCSA) in the leg of patients affected by mitochondrial diseases. The hypothesis is that there can be a disrupted relationship between strength and CCSA.

DETAILED DESCRIPTION:
Mitochondrial disorders are a group of inherited disorders caused by mutations in genes encoding mitochondrial proteins. The proteins are encoded by genes from both the mitochondrial DNA (mtDNA) and the nucleus, making some of the disorders maternally inherited and some autosomal recessive or dominant.

The mitochondria are found in almost all cells in the body and are the main source of energy. The energy is produced through the electron transport chain, which is composed of four multi subunit complexes (I to IV). A mutation in one or more of these complexes is a typical cause of a mitochondrial disease.

Since the mitochondria are found in almost every cell, mitochondrial disease can give rise to symptoms from many organs. The symptoms depend on what kind of mutation the patient has, but usually includes muscular and neurological problems, as these cells have especially high energy needs.

It is believed that the muscle weakness in mitochondrial diseases is caused by the reduced ability to produce energy. However, recent research has suggested that there is a structural change in the muscles as well. The hypothesis is that this structural change in the muscles will affect its function.

The aim of the study is to investigate the relation between muscle strength and contractile cross sectional area (CCSA) in the calf of patients affected by mitochondrial diseases. In healthy individuals there is a close relation between strength and CCSA, as the strength will decrease according to a decrease in CCSA. In mitochondrial disease, the hypothesis is that there can be a disrupted relationship between strength and CCSA.

The investigators will recruit 30 subjects with verified mitochondrial disease, and compare the results to that of healthy individuals (results from an earlier research project). A Dixon MRI will be used to find the CCSA of the calf muscle and a muscle dynamometer will be used to find the strength. These two variables are compared.

ELIGIBILITY:
Inclusion Criteria:

* Verified mitochondrial disease.
* Age: Over 18 years old

Exclusion Criteria:

* Contraindications for an MRI.
* Claustrophobia.
* Pregnant or nursing women.
* Competing disorders (as arthritis) or other muscle disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with verified mitochondrial disease.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2016-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Muscle CCSA, investigated by Dixon MRI techniques. | One MRI scan per subject (exam lasts approximately 60 min.)
  The MRI protocol include a whole body scan. The calf is chosen for qualitative analysis. Cross sectional area is calculated, the amount of adipose tissue is calculated, and the amount of adipose tissue is subtracted from the CSA, giving the CCSA.
Muscle strength, measured as peak torque, investigated by an isokinetic dynamometer (Biodex 4). | The tests takes less than an hour and are only done once.
  The dynamometer makes it possible to isolate particular muscle groups. It is possible to control the range of motion and thereby test in an area free of pain.

SECONDARY OUTCOMES:
Assessment of the muscle strength by a clinical test using "the Medical Research Council Scale for muscle strength" (MRC-scale). | The exam lasts 15 min.

CONTACTS AND LOCATIONS:
Overall Officials: Nanna S Nielsen, B.Sc, Principal Investigator — Copenhagen Neuromuscular Center
Locations (1):
- Rigshospitalet, Copenhagen, Copenhagen East, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lightowlers RN, Taylor RW, Turnbull DM. Mutations causing mitochondrial disease: What is new and what challenges remain? Science. 2015 Sep 25;349(6255):1494-9. doi: 10.1126/science.aac7516. Epub 2015 Sep 24. PMID 26404827
- [Background] Paternostro-Sluga T, Grim-Stieger M, Posch M, Schuhfried O, Vacariu G, Mittermaier C, Bittner C, Fialka-Moser V. Reliability and validity of the Medical Research Council (MRC) scale and a modified scale for testing muscle strength in patients with radial palsy. J Rehabil Med. 2008 Aug;40(8):665-71. doi: 10.2340/16501977-0235. PMID 19020701
- See also: Home page with knowledge about mitochondrial diseases. Used to write the "Background" in the study protocol. — http://www.mda.org/disease/mitochondrial-myopathies